CLINICAL TRIAL: NCT00676195
Title: An Open-Label Study of N-Acetyl Cysteine in Autism
Brief Title: An Open-Label Study of N-Acetyl Cysteine in Children With Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-05062008-1139
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Autistic Disorder
Keywords: N-Acetyl Cysteine
MeSH Terms: conditions — Autistic Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N-Acetyl Cysteine (Experimental): Dosage of orally administered N-Acetyl Cysteine is as follows:
  Days 1-30: 900 mg, once per day Days 31-60: 900 mg, twice per day Days 61-90: 900 mg, three times per day
  Interventions: Drug: N-Acetyl Cysteine

INTERVENTIONS:
Drug: N-Acetyl Cysteine — Dosage of orally administered N-Acetyl Cysteine is as follows:
  Days 1-30: 900 mg, once per day Days 31-60: 900 mg, twice per day Days 61-90: 900 mg, three times per day
  Other Names: NAC

SUMMARY:
The purpose of the study is to test the tolerability and efficacy of N-Acetyl Cysteine (NAC) in children with Autism.

DETAILED DESCRIPTION:
N-Acetyl Cysteine (NAC) is a compound that increases the levels of Glutathione, the body's main antioxidant. Glutathione is a compound in the blood that is part of a natural defense system (the antioxidant system). Anti-oxidants protect the body from damage caused by internal toxins called free radicals. It is possible that children with Autism tend to have lower levels of glutathione, an important compound in our bodies that helps combat the effects of toxic free radicals. We hope that by studying the antioxidant system in more detail, we will increase our understanding of the reasons why people develop Autism so that we can design better ways to treat individuals with this condition. This study is meant to test the safety tolerability of N-Acetyl Cysteine and its effectiveness in the treatment of behavioral difficulties in children with autism. It will also examine the possible benefit of this agent in improving the core deficits in autism such as social deficits.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for this study if they participated in the Double-blind, randomized, placebo controlled study of N-Acetyl Cysteine in Autism study at Stanford University and meet all of the following criteria:

1. Outpatients between 3.0 and 12.11 years of age inclusive
2. Males and females who are physically healthy
3. diagnosis of autism based on Diagnostic and Statistical Manual (DSM-IV-TR) criteria, the Autism Diagnostic Interview-Revised, and expert clinical evaluation
4. Clinical Global Impression Severity rating of 4
5. Care provider who can reliably bring subject to clinic visits, can provide trustworthy ratings, and interacts with subject on a regular basis
6. Ability of subject to swallow the compound
7. Stable concomitant medications for at least 2 weeks
8. No planned changes in psychosocial interventions during the open-label N-Acetyl Cysteine trial

Exclusion Criteria:

1. Diagnostic and Statistical Manual (DSM-IV-TR) diagnosis of schizophrenia, schizoaffective disorder, or psychotic disorder, not otherwise specified
2. Active medical problems: unstable seizures, significant physical illness (e.g., serious liver or renal pathology)
3. Pregnancy or sexually active females
4. Subjects taking antioxidant agents and glutathione prodrugs will be excluded from the study except if they have been off these compounds for at least 4 weeks

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-Acetyl Cysteine
Started | 24
Completed | 21
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | N-Acetyl Cysteine
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Reported on the Dosage Record and Treatment Emergent Symptom Scale (DOTES)
Description: Number of Participants with adverse events reported on the Dosage Record and Treatment Emergent Symptom Scale (DOTES) during the course of the study as measured at time points (4, 8, and 12 weeks).
Time Frame: 4, 8, and 12 weeks
Measure: Number; unit: number of participants
Arm/Group | N-Acetyl Cysteine
Number analyzed (Participants) | 24
number of participants | 17

2. Secondary Outcome: Social Responsiveness Scale (SRS)
Time Frame: 12 weeks
Population: No analyses were conducted since it is an open-label trial and data was analyzed in the double-blind phase. Additionally, the main reason for the this phase is to allow participants who were on the placebo during the double-blind phase of NCT00627705 to receive the compound.
Arm/Group | Open-Label
Number analyzed (Participants) | 0

3. Secondary Outcome: Sensory Profile Questionnaire (SPQ)
Time Frame: 12 weeks
Population: as for outcome 2
Arm/Group | Open-Label
Number analyzed (Participants) | 0

4. Secondary Outcome: Irritability Subscale of the Aberrant Behavior Checklist (ABC)
Time Frame: 4, 8, and 12 weeks
Population: as for outcome 2
Arm/Group | Open-Label
Number analyzed (Participants) | 0

5. Secondary Outcome: Glutathione Metabolism Intermediates in Peripheral Blood Measured by High-performance Liquid Chromatography
Time Frame: 12 weeks
Population: as for outcome 2
Arm/Group | Open-Label
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline and 4, 8 and 12 Weeks.
Arm/Group | N-Acetyl Cysteine
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 19/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetyl Cysteine (N=24)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Decreased Appetite (Gastrointestinal disorders) | 5 (6)
Depressive Affect (Psychiatric disorders) | 3 (3)
Nasal Congestion (General disorders) | 6 (6)
Insomnia (General disorders) | 4 (4)
Decreased Motor Activity (General disorders) | 2 (2)
Grinding Teeth (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This is an open-label trial with a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No